CLINICAL TRIAL: NCT03217305
Title: NAVA vs Pressure Support After Cardiac Surgery, a Physiological Study
Brief Title: Neurally Adjusted Ventilatory Assist (NAVA) vs Pressure Support Ventilation After Cardiac Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Martinsson, MD, Göteborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMartinssonthorax2
Record Dates: First submitted 2017-06-21; First posted 2017-07-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Ventilator Lung
Keywords: EIT. NAVA. Endexpiratory Lung Impedance.

STUDY DESIGN:
Intervention Model Description: Control-Intervention-Control
Masking Description: The investigator works as physician at the Department of Intensive Care. The participants are patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAVA vs Pressure Support (Other): Control (pressure support) - NAVA - Control (Pressure Support) Intervention is NAVA
  Interventions: Device: NAVA

INTERVENTIONS:
Device: NAVA — Neurally Adjusted Ventilatory Assist is a fairly new ventilation mode

SUMMARY:
The study compares two different ventilation modes, Pressure support ventilation vs. Neuronally Adjusted Ventilatory Assist, in postcardiac surgery patients. Of special interest is shunt and alveolar deadspace and ventral vs. dorsal ventilation.

DETAILED DESCRIPTION:
The aim of the study is to compare two different ventilation modes in complicated postcardiac surgery patients, who need ventilatory support during weaning phase, in the Cardiothoracic Intensive Care Unit. The two different ventilation modes are Neuronally Adjusted Ventilatory Assist (NAVA) and Pressure Support ventilation. NAVA ventilation mode have been introduced a couple of years ago as an alternative to pressure support. The advantage of NAVA mode compared to pressure support is a better synchrony between patient and ventilator in the inspired and expired phases. Maybe there are also physiological advantages of the NAVA mode, which we want to study in the present study.

All patients have three measurement periods. 1) Pressure support during 20 min, NAVA equilibration period of 30 min, followed by 2) NAVA ventilation for 20 min, pressure support equilibration period of 30 min and 3) pressure support for 20 min. Blood gases and cardiac output measurements is performed before and after each measurement period. Regional ventilation is measured by Electric Impedance Tomography (EIT).

ELIGIBILITY:
Inclusion Criteria:

* Complicated Post Cardiac surgery patients in the ventilator weaning phase.
* Patients requiring assisted ventilation
* Respiratory and circulatory stable patients
* Sedated patients, RASS -2 to -3

Exclusion Criteria:

* Transplanted patients
* Pleural effusion.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Ventilation distribution | Through study completion, within approximately 18 months
  Redistribution of ventilation , dorsally vs. ventrally
Alveolar dead space | Through study completion, within approximately 18 months
  Calculated from blood gases and end tidal pCO2,using standard formulae
End expiratory lung impedance | Through study completion, within approximately 18 months
  Measured by Electric Impedance Tomography
PaO2/FiO2 | Through study completion, within approximately 18 months
  Arterial oxygenation
Alveolar shunt | Through study completion, within approximately 18 months
  Calculated from mixed venous and arterial blood gases

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thoren, MD, PhD, Principal Investigator — University of Goteborg
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinsson A, Lundholm C, Ricksten SE, Oras J, Magnusson JM, Wallinder A, Sellgren J, Thoren A. Neurally adjusted ventilatory assist vs pressure support ventilation: short-term effects on shunt and dead space after cardiac surgery. Sci Rep. 2025 Dec 21;15(1):44234. doi: 10.1038/s41598-025-33097-1. PMID 41423634